CLINICAL TRIAL: NCT05924100
Title: Efficacy and Safety of Luspatercept for the Treatment of Anemia Due to Myelodysplastic Syndromes With del5q, Refractory/Resistant/Intolerant to Prior Treatments, Who Require Red Blood Cell Transfusions
Brief Title: Efficacy and Safety of Luspatercept for the Treatment of Anemia Due to MDS With del5q, Refractory/Resistant/Intolerant to Prior Treatments, RBC-TD
Acronym: Phoenix
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Associazione Qol-one (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QOL-ONE Phoenix
Record Dates: First submitted 2023-06-08; First posted 2023-06-29 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Myelodysplastic Syndromes; Del(5Q); Anemia; Transfusion-dependent Anemia
Keywords: MDS with Del(5Q)
MeSH Terms: conditions — Myelodysplastic Syndromes; Anemia | interventions — luspatercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Luspatercept (Experimental)
  Interventions: Drug: Luspatercept Injection [Reblozyl]

INTERVENTIONS:
Drug: Luspatercept Injection [Reblozyl] — Eligible subjects will receive luspatercept (ACE-536): starting dose of 1.0 mg/kg subcutaneous injection every 3 weeks (21 days; Q3W). Dose levels can be increased in a stepwise manner beyond the starting dose to 1.33 mg/kg, and up to a maximum of 1.75 mg/kg (with a maximum total dose of 168 mg).
  All subjects who have received at least one dose of luspatercept should undergo follow-up evaluations after day 169 with Assessment visits every 24 weeks (168 days) up to 2 years to evaluate evidence of clinical benefit.

SUMMARY:
Myelodysplastic syndromes, primarily affecting older adults, are a heterogeneous group of clonal disorders of hematopoietic stem cells characterized by ineffective hematopoiesis that manifest clinically as anemia, neutropenia, and/or thrombocytopenia of variable severity; these often result in RBC- transfusion dependent (TD) anemia, increased risk of infection, and/or hemorrhage, as well as a potential to progress to acute myeloid leukemia (AML).

Lenalidomide is approved for red blood cell transfusion-dependent (RBC TD) anemia due to low-risk myelodysplastic syndromes (MDS) with a chromosome 5q deletion (del5q) with or without additional cytogenetic abnormalities. About one third of patients are refractory/resistant/intolerant and will require further treatment options.

Luspatercept (ACE-536), an erythroid maturation agent, is a recombinant fusion protein consisting of a modified form of the extracellular domain (ECD) of the human activin receptor type IIB (ActRIIB) linked to the Fc portion of human immunoglobulin G1 (IgG1-Fc). Luspatercept acts on endogenous inhibitors of late-stage erythropoiesis (eg, growth differentiation factor 11, GDF11) to increase release of mature erythrocytes into circulation. Nonclinical data have demonstrated that luspatercept binds to negative regulators governing late-stage erythroid development to inhibit their action, thereby promoting the maturation of erythrocytes in the bone marrow.

Luspatercept is indicated for the treatment of adult patients with transfusion-dependent anaemia associated with beta-thalassaemia and due to very low, low and intermediate-risk MDS with ring sideroblasts, who had an unsatisfactory response to or are ineligible for erythropoietin-based-therapy. It is not indicated for other MDS subtypes. Unfortunately, patients with MDS with del5q refractory/resistant/intolerant to lenalidomide are excluded from clinical trials that evaluate novel treatments for the anemia of RBC TD lower risk MDS. Therefore, treatment of anemia in such patients is an unmet need.

QOL-ONE Phoenix is a Phase 2, multicenter, single arm, prospective study. The primary objective of the study is to evaluate the effect of luspatercept on RBC TI in subjects with MDS with del5q with IPSS-R very low, low, or intermediate risk and < 5% bone marrow blasts, resistant/refractory/intolerant to lenalidomide and who require RBC transfusions.

The study is divided into a Screening Period, a 2-year Treatment Period and a 3-year Follow-up Period.

Primary objective is to evaluate the effect of luspatercept on RBC TI (lack of transfusions for 8 consecutive weeks within the first 24 weeks) in subjects with MDS with del5q with IPSS-R very low, low, or intermediate risk and < 5% bone marrow blasts, resistant/refractory/intolerant to lenalidomide and RBC TD.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must understand and voluntarily sign an ICF prior to any study-related assessments/procedures being conducted.
2. Documented diagnosis of MDS with del5q according to 2018 WHO classification
3. IPSS-R classification (Greenberg, 2012) of very low, low, or intermediate risk disease, and:

   * < 5% blasts in bone marrow
   * Peripheral blood WBC count <13,000/μL
4. Refractory or intolerant to, or ineligible for, prior ESA treatment
5. If previously treated with ESAs or granulocyte colony-stimulating factor (G-CSF), both agents must have been discontinued ≥ 4 weeks prior to date of screening.
6. Refractory or intolerant to, or ineligible for, prior lenalidomide treatment, as defined by any one of the following:

   * Refractory to prior lenalidomide treatment for at least 4 cycles; - documentation of non-response or response that is no longer maintained (HI-E)
   * Intolerant to prior lenalidomide treatment - documentation of discontinuation of lenalidomide at any time after introduction due to intolerance or an adverse event
   * lenalidomide ineligible -platelet counts below 50000/mmc or absolute neutrophil count below 500/mmc at the start of treatment
   * lenalidomide must have been discontinued ≥ 4 weeks prior to date of screening.

   Requires RBC transfusions, as documented by the following criteria:
   * average transfusion requirement of ≥ 2 units/8 weeks of pRBCs confirmed for a minimum of 16 weeks immediately preceding enrolment.
   * Hb levels at the time of or within 7 days prior to administration of a RBC transfusion must have been ≤ 10.0 g/dL in order for the transfusion to be counted towards meeting eligibility criteria. RBC transfusions administered when Hb levels were > 10.0 g/dL and/or RBC transfusions administered for elective surgery will not qualify as a required transfusion for the purpose of meeting eligibility criteria.
   * no consecutive 56-day period that was RBC transfusion-free during the 16 weeks immediately preceding screening
7. Eastern Cooperative Oncology Group (ECOG) score of 0, 1, or 2
8. Females of childbearing potential, defined as a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy or 2) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (ie, has had menses at any time in the preceding 24 consecutive months), must:

   * Have two negative pregnancy tests as verified by the Investigator prior to starting study therapy (unless the screening pregnancy test was done within 72 hours of C1D1). Refer to Section 6.1 for additional details. She must agree to ongoing pregnancy testing during the course of the study, and after the end of study treatment.
   * If sexually active, agree to use, and be able to comply with, highly effective contraception without interruption, 5 weeks prior to starting investigational product, during the study therapy (including dose interruptions), and for 12 weeks after discontinuation of study therapy.
9. Male subjects must:

   * Agree to use a condom, defined as a male latex condom or non latex condom not made out of natural (animal) membrane (for example, polyurethane), during sexual contact with a pregnant female or a female of childbearing potential while participating in the study, during dose interruptions and for at least 12 weeks following investigational product discontinuation, even if he has undergone a successful vasectomy.
10. Subject is willing and able to adhere to the study visit schedule and other protocol requirements.

Exclusion Criteria:

1. P53 mutation at screening
2. Prior therapy with disease modifying agents for underlying MDS disease (hypomethylating agents)

   * subjects who previously received HMA may be enrolled at the investigator's discretion contingent that the subject received no more than 1 dose of HMA). The last dose must be ≥ 5 weeks from the date of screening.
3. Previously treated with either luspatercept (ACE-536) or sotatercept (ACE-011)
4. Secondary MDS, ie, MDS that is known to have arisen as the result of chemical injury or treatment with chemotherapy and/or radiation for other diseases. 5 Known clinically significant anemia due to iron, vitamin B12, or folate deficiencies, or autoimmune or hereditary hemolytic anemia, or gastrointestinal bleeding

6. Prior allogeneic or autologous stem cell transplant 7. Known history of diagnosis of AML 8. Use of any of the following within 5 weeks prior to study entry:

* anticancer cytotoxic chemotherapeutic agent or treatment
* corticosteroid, except for subjects on a stable or decreasing dose for ≥ 1 week prior to study entry for medical conditions other than MDS
* iron-chelating agents, except for subjects on a stable or decreasing dose for at least 8 weeks prior to screening
* other RBC hematopoietic growth factors
* investigational drug or device, or approved therapy for investigational use. If the half- life of the previous investigational product is known, use within 5 times the half- life prior to screening or within 5 weeks, whichever is longer is excluded. 9. Uncontrolled hypertension, defined as repeated elevations of diastolic blood pressure (DBP) ≥ 100 mmHg despite adequate treatment. 10. Estimated glomerular filtration rate (eGFR) or creatinine clearance < 40 mL/min.

  11. Serum aspartate aminotransferase/serum glutamic oxaloacetic transaminase or alanine aminotransferase/serum glutamic pyruvic transaminase ≥ 3.0 x upper limit of normal (ULN) 12. Total bilirubin ≥ 2.0 x ULN.
* higher levels are acceptable if these can be attributed to active red blood cell precursor destruction within the bone marrow (ie, ineffective erythropoiesis) or in the presence of known history of Gilbert Syndrome.
* subjects are excluded if there is evidence of autoimmune hemolytic anemia 13. Prior history of malignancies, other than MDS, unless the subject has been free of the disease (including completion of any active or adjuvant treatment for prior malignancy) for ≥ 5 years. However, subjects with the following history/concurrent conditions are allowed:
* Basal or squamous cell carcinoma of the skin
* Carcinoma in situ of the cervix
* Carcinoma in situ of the breast
* Incidental histologic finding of prostate cancer (T1a or T1b using the tumor, nodes, metastasis [TNM] clinical staging system)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2022-11-03 (Actual); Primary Completion 2024-12-03 (Estimated); Study Completion 2029-12-03 (Estimated)

PRIMARY OUTCOMES:
RBC Transfusion Independence | 24 WEEKS
  Proportion of subjects who are RBC TI for 8 weeks over the first 24 weeks from trial entry

SECONDARY OUTCOMES:
Safety and tolerability of Luspatercept measured as frequency and severity of adverse events occurred and assessed by CTCAE v. 5.0 | 5 years
  Type, frequency, severity of AEs. The adverse events occurring in the subjects enrolled in the study will be evaluated according to CTCAE v5.0 Furthermore, the relationship between adverse events and treatment with luspatercept will be evaluated
RBC-TI in long term | 5 years
  Proportion of subjects who are RBC TI for 8 weeks over the first 48 weeks from trial entry and over the 30 months
Duration of RBC-TI | 2 years
  Maximum duration of RBC transfusion independence for subjects who achieve RBC TI ≥ 8 weeks
Reduction in RBC transfusions | 24 weeks
  Mean change in total pRBC units transfused over a rolling 8-week period and proportion achievieng HI-E (reduction in ≥ 4 units in the preceding 8 weeks in those with baseline transfusion burden of ≥8 units in 8 preceding weeks)
Increase in hemoglobin | 2 years
  Mean change in hb levels from baseline and proportion achieving HI-E (gain in Hb ≥1.5 g/dL)
Change in quality of life scores with QOL-E questionnaire | 2 years
  Scores of QOL-E questionnaire from baseline and proportion achieving meaningful clinical important difference). Higher values indicate better quality of life
Change in quality of life scores with HM-PRO questionnaire | 2 years
  Scores of HM-PRO questionnaire from baseline and proportion achieving meaningful clinical important difference). Lower values indicate better quality of life
Change in Serum Ferritin | 2 years
  Mean change of the value of serum ferritin from baseline.
Change in iron chelation therapy use | 2 years
  Mean change of dose of iron chelation therapy use from baseline
Time to RBC TI | 2 years
  Time to achieving first RBC TI ≥ 8 weeks in the first 24 weeks

CONTACTS AND LOCATIONS:
Locations (23):
- Italy (23):
  - A.O. SS. Antonio e Biagio e Cesare Arrigo Ospedale Civile, Alessandria
  - A.O.U. Ospedali Riuniti, Ancona
  - A.O. S. Giuseppe Moscati, Avellino
  - Ospedale degli Infermi, Biella
  - A.O.U. G. Rodolico San Marco, Catania
  - ARNAS Garibaldi, PO Nesima, Catania
  - ASL TO 4 - Ospedale Chivasso, Chivasso
  - Azienda Ospedaliera Annunziata, Cosenza
  - A.O.U. Careggi, Florence
  - A.O.U. Federico II, Napoli
  - A.O.U. Maggiore della Carità, Novara
  - A.O.U. Policlinico Paolo Giaccone, Palermo
  - Ospedale Civile Spirito Santo, Pescara
  - Grande Ospedale Metropolitano Bianchi-Melacrino-Morelli, Reggio Calabria
  - IRCCS di Reggio Emilia, Reggio Emilia
  - Ospedale S. Eugenio, Roma
  - Policlinico Tor Vergata, Roma
  - Policlinico Umberto I, Roma
  - A.O.U. San Giovanni di Dio e Ruggì D'Aragona, Salerno
  - Casa Sollievo della Sofferenza IRCCS, San Giovanni Rotondo
  - AO Santa Maria di Terni, Terni
  - A.O. Città della Salute e della Scienza, Torino
  - ASU Giuliano Isontina, Trieste